CLINICAL TRIAL: NCT06373133
Title: An Exploratory Clinical Trial of SHR-8068 Combined With Aldebelizumab and BP102 in the Treatment of Refractory Colorectal Cancer
Brief Title: SHR-8068 Combined With Adbelizumab and BP102 in the Treatment of Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dan Cao, Chief physician, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024 (82)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-8068+Adebrelimab+BP102 (Experimental): The first 9 subjects will be treated with low dose SHR-8068 (1mg/kg, q6w), and the subsequent subjects will be treated with high dose SHR-8068 (4mg/kg, q12w) if the toxicity of DLT is tolerable during the observation period.
  Interventions: Drug: SHR-8068; Drug: Adebrelimab; Drug: BP102

INTERVENTIONS:
Drug: SHR-8068 — 1mg/kg，ivgtt, d1, q6w or 4mg/kg，ivgtt, d1, q12w
  Other Names: Anti-CTLA4 monoclonal antibody
Drug: Adebrelimab — 1200mg, ivgtt, d1, q3w
  Other Names: SHR-1316
Drug: BP102 — 7.5mg/kg, ivgtt, d1, q3w
  Other Names: Bevacizumab

SUMMARY:
To evaluate the efficacy and safety of SHR-8068 and Adebrelimab in Combination With Bevacizumabin in the treatment of microsatellite stable (MSS) advanced colorectal cancer.

DETAILED DESCRIPTION:
Previous studies have found that PD-1 or PD-L1 inhibitors combined with CTLA-4 inhibitors have better efficacy than PD-1 or PD-L1 inhibitors alone. Anti-angiogenesis targeted drugs can enhance the anti-tumor effects of immune checkpoint inhibitors by reducing the activity of immunosuppressive cells and normalizing tumor vascular structure, and its combination with immunotherapy has become a standard regimen in liver cancer. Based on the above, this study aims to explore the efficacy and safety of SHR-8068 and adbelizumab combined with bevacizumab in the treatment of MSS type of metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed metastatic colorectal adenocarcinoma;
2. Age of 18-75 years old, both sexes;
3. predicted survival time ≥12 weeks;
4. Eastern Cooperative Oncology Group performance status (ECOG) score 0-2;
5. Participants who had failed second-line or higher standard-of-care systemic therapy and should have been treated with oxaliplatin, irinotecan, and fluorouracil were allowed to enroll if first-line therapy included three agents;
6. liver tumor burden ≤50% as assessed by enhanced CT or MRI;
7. There were no serious complications (perforation, obstruction, massive bleeding, etc.) in the primary lesion;
8. According to RECIST1.1 criteria, there should be at least one measurable objective tumor lesion, the maximum diameter of which must be ≥1cm by spiral CT, and the maximum diameter of which must be ≥2cm by conventional CT or MRI; This procedure was performed within 28 days before enrollment.
9. Study participants had to have adequate organ function, as assessed by the following laboratory results within 1 week before enrollment (no blood transfusion, granulocyte colony-stimulating factor, or other medical support within 14 days before study drug administration) :

   1. Blood routine examination: hemoglobin ≥90g/L; Platelet (PLT) ≥75×109/L; White blood cell (WBC) ≥3.0×109/L; Neutrophil (ANC) ≥1.5×109/L;
   2. Blood biochemical examination: total bilirubin (TBI) ≤1.5× upper limit of normal (UNL); Serum creatinine (Cr) ≤1.5× upper limit of normal; Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤5×UNL;
10. study participants with active hepatitis B or active hepatitis C, who must have received antiviral therapy for at least 14 days before the first dose of the study drug, If they have a hepatitis B virus (HBV) DNA titer test (not higher than 500 IU/mL or 2500 copies [cps]/mL) and a hepatitis C virus (HCV) RNA test (not higher than the lower limit of detection of the assay), can be enrolled in the trial, and are willing to continue to receive effective antiviral therapy during the study;
11. Patients volunteered to participate and provided written informed consent.

Exclusion Criteria:

1. a history of other malignancies with disease-free survival <5 years (except cured basal cell carcinoma of the skin, cured carcinoma in situ of the cervix, and gastrointestinal cancer proven cured by endoscopic mucosal resection);
2. participated in other drug clinical trials within four weeks;
3. patients with known CNS metastases or a history of CNS metastases before screening. For patients with clinically suspected central nervous system metastasis, contrast-enhanced CT or contrast-enhanced magnetic resonance imaging (MRI) was required within 28 days before informed consent to rule out central nervous system metastasis.
4. patients with a long history of chronic diarrhea or complete intestinal obstruction;
5. urinalysis showed urinary protein ≥2+ or 24-hour urinary protein ≥1g;
6. Drug-uncontrolled hypertension (systolic blood pressure > 140 MMHG or diastolic blood pressure > 90mmHg);
7. a history of severe bleeding (> 30ml per episode) within 3 months or hemoptysis (> 5ml per episode) within 1 month or thromboembolic events (including pulmonary embolism, cerebral infarction, etc.) within 12 months;
8. had undergone surgical treatment (excluding biopsy) within 6 weeks or had unhealed surgical incisions;
9. long-term unhealed wounds or incompletely healed fractures;
10. imaging shows that the tumor has invaded the vital blood vessels or the patient's tumor has a high possibility of invading the vital blood vessels during treatment, which may cause fatal bleeding;
11. with a history of unstable angina pectoris; Newly diagnosed angina pectoris within 3 months before screening or myocardial infarction within 6 months before screening; Arrhythmias (including QTcF ≥450 ms in men and ≥470 ms in women) required long-term use of antiarrhythmic drugs and New York Heart Association (NYHA) grade ≥II cardiac dysfunction.
12. patients with abnormal coagulation function and bleeding tendency (INR within the normal range without anticoagulant therapy must be met within 14 days before the first medication); Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogues; Low-dose warfarin (1 mg orally once daily) or low-dose aspirin (at a dose of up to 100 mg daily) for preventive purposes were allowed if the International Normalized Ratio of prothrombin time (INR) was 1.5 or less.
13. participants with an active or prior autoimmune disease or risk (e.g., organ transplant requiring immunosuppressive therapy) that may relapse. However, participants with type 1 diabetes, hypothyroidism for which they were receiving hormone-replacement therapy only, or skin conditions for which no systemic treatment was required (e.g., vitiligo, psoriasis, or alopecia) were allowed.
14. have had a history of interstitial lung disease or noninfectious pneumonia, such as symptomatic disease or a previous pulmonary history that may preclude assessment or management of study-drug-related pulmonary toxicity;
15. Participants with a history of active pulmonary tuberculosis infection within 1 year before the first dose of the study drug and a history of active pulmonary tuberculosis infection more than 1 year before were considered eligible if they had no evidence of current active pulmonary tuberculosis, as assessed by the investigator;
16. severe uncontrolled medical illness or acute infection (fever > 38 ° C);
17. study participants who required systemic treatment with corticosteroids (>10 mg/ day prednisone equivalent dose) or other immunosuppressive drugs within 14 days prior to administration of the study drug. Note: In the absence of active autoimmune disease, inhaled or topical steroid hormones, or adrenal hormone replacement therapy with an equivalent dose of ≤10 mg prednisone per day, were allowed. Short-term (≤ 7 days) use of glucocorticoids was permitted for preventive treatment (e.g., contrast allergy) or for the treatment of nonautoimmune conditions (e.g., delayed hypersensitivity from a contact allergen).
18. study participants who had been treated with any antibody/drug (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4, anti-OX-40, anti-CD137, anti-TIM-3, anti-LAG-3 antibodies, etc.) targeting a T-cell co-regulatory protein (immune checkpoint);
19. study participants with a history of allergic or hypersensitivity reactions to study drug components;
20. have immunodeficiency diseases or HIV infection;
21. pregnant or lactating women or patients of childbearing potential (men or women who have been without menstruation for less than 1 year) who are unwilling to use contraception;
22. concomitant diseases that, according to the investigator's judgment, seriously endanger the patient's safety or prevent the patient from completing the study;
23. who were deemed by the investigator to be ineligible for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | The first 21 days of the first cycle of medication
  The dose is considered tolerable if the incidence of DLT is less than 33.3%.
PFS | Up to 2 years
  Progression-free survival (PFS) denotes the chances of staying free of disease progression for a group of individuals suffering from a cancer after a particular treatment.